CLINICAL TRIAL: NCT03232892
Title: Phase II Trial to Evaluate Trametinib in Patients With Advanced NF1-mutant Non-small Cell Lung Cancer
Brief Title: Trametinib in Patients With Advanced Neurofibromatosis Type 1 (NF1)-Mutant Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 166521; NCI-2017-02295 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-07-14; First posted 2017-07-28 (Actual); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; NF-1 mutant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trametinib

STUDY DESIGN:
Intervention Model Description: Phase 2, single-arm, open label, multicenter clinical trial.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trametinib 2.0mg PO daily (Experimental): Trametinib 2.0mg PO daily in 28-day cycles. A maximum of two trametinib dose level reductions are allowed (1.5mg and 1mg) in the case of adverse reactions.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — Trametinib 2mg, once daily, PO, 28-day cycles
  Other Names: Mekinist

SUMMARY:
Phase II trial to evaluate trametinib in patients with locally advanced non-squamous, non-small cell lung cancer (NSCLC) whose tumors harbor a non-synonymous NF-1 mutation, with progressive disease on at least one prior line of therapy.

DETAILED DESCRIPTION:
This is a phase II, single-arm, open-label, multicenter clinical trial evaluating the efficacy and safety of trametinib monotherapy in patients with advanced non-squamous NSCLC whose tumors non-synonymous NF1 mutations and are KRAS wildtype. Eligible patients must have documented disease progression either during or after treatment with most recent therapy and may not have received prior treatment with a MEK inhibitor. Patients with activating alterations in EGFR, ALK, and ROS-1 must also have received appropriate TKI treatment. Patients who meet eligibility criteria will receive trametinib monotherapy and followed for the primary endpoint of objective response rate and additional secondary endpoints. A total of 27 patients will be enrolled into the study, with the goals of obtaining 24 evaluable patients. Patients may continue treatment until disease progression or up to 24 months from the time of study entry or until the study is closed. All patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or unresectable locally advanced, non-squamous, NSCLC.
2. Documented non-synonymous somatic mutation in NF1 in any tumor specimen or cell-free DNA assay by Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory.
3. Received at least one prior line of cancer therapy for the treatment of NSCLC; this should include at least one of the following: platinum (carboplatin or cisplatin) doublet chemotherapy (acceptable combinations include: paclitaxel, docetaxel, abraxane, pemetrexed, gemcitabine, vinorelbine, or etoposide), anti-PD1/PDL1 therapy (pembrolizumab, nivolumab, or atezolizumab), or appropriate targeted therapy in patients with activating EGFR (osimertinib, erlotinib, gefitinib, or afatinib), ALK (alectinib, crizotinib, ceritinib, brigatinib, or loralatinib), or ROS-1 (crizotininb or entrectinib) alterations; therapy may be given as monotherapy or in combination with other cancer therapy (e.g. bevacizumab, ipilumimab)
4. Patients with a known activating mutation in epidermal growth factor receptor (EGFR) (Exon 19 deletion, G719A, S768I, V769L, T790M, L833F, L858R, L861Q), must have progressed or been intolerant to treatment with a first-line EGFR tyrosine kinase inhibitor (TKI) (erlotinib, afatinib, or gefitinib). Patients whose tumors were found to have an EGFR T790M mutation must also have progressed or been intolerable to treatment with osimertinib.
5. Patients with a known Anaplastic lymphoma kinase (ALK)-rearrangement must have progressed or been intolerant to treatment with at least one ALK TKI: crizotinib ceritinib, alectinib,brigatinib, or loralatinib
6. Patients with a known ROS-1-rearrangement must have progressed or been intolerant to treatment with crizotinib or entrectinib
7. Patients with PDL1 level of >= 50%, who do not have an ALK-rearrangement or EGFR-mutation, must have progressed or been intolerant to treatment with anti-PD1/PDL1 therapy (pembrolizumab, nivolumab, or atezolizumab)
8. Documented disease progression or intolerance to treatment either during or after treatment with most recent therapy.
9. Willingness to undergo research biopsy.
10. Measurable disease defined by RECIST 1.1 criteria.
11. Life expectancy of at least 3 months.
12. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
13. Age ≥ 18 years.
14. Resolution of all acute toxic effects of prior chemotherapy, immunotherapy, radiotherapy or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 grade 1.
15. Adequate baseline organ function defined as follows:

    Hematologic:
    * Absolute neutrophil count: ≥ 1.2 x 10^9/L
    * Hemoglobin: ≥ 9 g/dL
    * Platelets: ≥ 100 x 10^9/L
    * PT/INR and PTT: ≤ 1.5 x upper limit of normal (ULN)

    Hepatic:
    * Albumin: ≥ 2.5 g/dL
    * Total bilirubin: ≤ 1.5 x ULN
    * AST and ALT: ≤ 2.5 x ULN

    Renal:
    * Creatine: ≤ 1.5 ULN or
    * Calculated creatinine clearance (calculated by the Cockcroft-Gault formula): ≥ 50 mL/min

    Cardiac:

    - Left Ventricular Ejection Fraction (LVEF): ≥ lower limit of normal (LLN) by echocardiogram (ECHO) or multiple-gated acquisition (MUGA)
16. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to study enrollment. The effects of trametinib on the developing human fetus are unknown. For this reason and because animal studies with trametinib have shown reproductive toxicity, women of child-bearing potential and men must agree to use effective methods of contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and for 4 months following discontinuation of trametinib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study drug administration.
17. Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
18. All prior treatment- related toxicities must be CTCAE (Version 4.03) ≤ Grade 1 (except alopecia) at the time of randomization
19. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Known mutation in KRAS at position G12, G13, or Q61.
2. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Treated brain metastases are allowed as long as they are stable for at least 28 days post-treatment.
3. Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with trametinib . Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with trametinib, breastfeeding should be discontinued if the mother is treated with trametinib.
4. History of another malignancy. Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer and/or subjects with indolent second malignancies are eligible.
5. Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
6. The subject has received cytotoxic chemotherapy, molecular targeted therapy, or immunotherapy within 21 days before the first dose of study drug (trametinib).
7. Prior treatment with MEK inhibitor.
8. History of interstitial lung disease or pneumonitis.
9. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
10. Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to study enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to study enrollment.
11. History of retinal vein occlusion (RVO).
12. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
13. History or evidence of cardiovascular risk including any of the following:

    * LVEF < LLN
    * A QT interval corrected for heart rate using the Bazett's formula (QTcB) ≥ 480 msec;
    * History or evidence of current clinically significant uncontrolled arrhythmias.
    * Clarification: Subjects with atrial fibrillation controlled (defined as not requiring change in cardiac drug dosing, emergency room visit, or hospital admission) for > 30 days prior to dosing are eligible.
    * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study enrollment.
    * History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association (NYHA).
    * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy;
    * Patients with intra-cardiac defibrillators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collin Blakely, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trametinib 2.0mg PO Daily
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was closed due to low accrual with a total of 1 participant enrolled on this protocol.
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  60-69 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: For participants receiving at least one dose of study treatment, the ORR is defined as the best overall response recorded from the start of the treatment until disease progression or recurrence as assessed over a 1-year period from the start of treatment. The frequency and percentages of patients with a best overall response rate of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be determined. We will test the hypothesis that the ORR is greater than the null hypothesis of 10% using the Fisher's exact test.
Time Frame: Up to 1 year
Population: The single participant did not allow for a sufficient data collection of endpoint analysis
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response (DR)
Description: The DR for Complete Response (CR) and Partial Response (PR) will be measured from the date that the best response is first recorded until the date that PD is documented. For patients who continue treatment post progression, the date of Disease Progression (PD) documentation will be used for analysis. The DR will be summarized using descriptive statistics (N, mean, standard deviation, minimum, and maximum).
Time Frame: Up to 4 years
Population: The single participant did not allow for a sufficient data collection of endpoint analysis
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate (DCR) According to RECIST Version 1.1 Criteria.
Description: DCR will be defined as the percentage of patients who have achieved CR, PR, or SD for at least 12 weeks. The DCR will be summarized using descriptive statistics (N, mean, standard deviation, minimum, and maximum).
Time Frame: Up to 4 years
Population: The single participant did not allow for a sufficient data collection of endpoint analysis
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 Criteria.
Description: PFS will be calculated as 1+ the number of days from the first dose of study drugs to documented radiographic progression or death due to any cause over a period of 1 year. For patients who continue treatment post-progression, the date of radiographic progression will be used for PFS analysis. For patients who continue treatment post-progression, the date of radiographic progression will be used for PFS analysis. The Kaplan-Meier analysis will be used to calculate the median PFS with 95% confidence interval.
Time Frame: Up to 1 year
Population: The single participant did not allow for a sufficient data collection of endpoint analysis
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS will be calculated as 1+ the number of days from the first dose of study drugs to death due to any cause over a period of 1 year. The Kaplan-Meier analysis will be used to calculate the median OS with 95% confidence interval.
Time Frame: Up to 1 year
Population: The single participant did not allow for a sufficient data collection of endpoint analysis
Arm/Group | Trametinib 2.0mg PO Daily
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: The safety population will consist of all subjects who receive any amount of study treatment which for this protocol is a total of 1 participant. Adverse event terms recorded on the CRFs were be mapped to preferred terms using the Medical Dictionary for Regulatory Activities (MedDRA). Seriousness, severity grade and relationship to study treatment will be assessed by the investigator. Severity grade will be defined by the National Cancer Institute (NCI) CTCAE v4.03
Arm/Group | Trametinib 2.0mg PO Daily
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trametinib 2.0mg PO Daily (N=1)
shortness of breath (Cardiac disorders) | 1 (1)
hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trametinib 2.0mg PO Daily (N=1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There was only one participant enrolled on this trial and the study was terminated early due to low accrual. No analyses were conducted on any of the samples collected as there was insufficient material available for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03232892/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03232892/Prot_SAP_001.pdf